CLINICAL TRIAL: NCT06366295
Title: Subgingival Mechanotherapy Using a Periodontal Endoscope Compared to Classical Subgingival Mechanotherapy for the Treatment of Periodontitis: a Randomized Clinical Trial
Brief Title: Comparison of Subgingival Mechanotherapy With and Without the Use of a Perioscope: Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WUM.Perio.05
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-06

CONDITIONS: Periodontitis
Keywords: periodontal endoscopy, perioscopy
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subgingival mechanotherapy with perioscopy (Experimental): Scaling and root planing using ultrasonic scaler and curettes, under the control of a perioscope, enabling real-time, magnified imaging of the root surface.
  Interventions: Device: subgingival mechanotherapy with perioscopy
- Classical subgingival mechanotherapy (Active Comparator): Scaling and root planing using ultrasonic scaler and curettes.
  Interventions: Device: classical subgingival mechanotherapy

INTERVENTIONS:
Device: subgingival mechanotherapy with perioscopy — Subgingival mechanotherapy using a machine scaler, curettes and a perioscope
  Arms: Subgingival mechanotherapy with perioscopy
Device: classical subgingival mechanotherapy — Subgingival mechanotherapy using a machine scaler and curettes
  Arms: Classical subgingival mechanotherapy

SUMMARY:
The study aims to comparatively assess clinical parameters, biochemical and microbiological parameters after treatment of periodontitis using subgingival mechanotherapy traditional and subgingival mechanotherapy using a perioscope.

DETAILED DESCRIPTION:
Non-surgical treatment is the basic form of disease treatment periodontitis. Its first stage is the mechanical removal of dental plaque along with the control of risk factors. Subgingival mechanotherapy, also known as scaling and root planing (SRP) is the next stage, aimed at the subgingival area. Perioscopy makes possible direct real-time visualization of the root surface during the procedure. The research results published so far indicate improvement or no significant differences clinical parameters after SRP procedure using a perioscope vs traditional subgingival instrumentation. The aim of this study is to indicate, or not, clinical, biochemical (level of pro-inflammatory cytokines) and microbiological (A. actinomycetemcomitans, P. gingivalis, T. denticola) differences after periodontitis treatment using the traditional method vs. using a perioscope.

ELIGIBILITY:
Inclusion Criteria:

* age 20-60; (II)
* preserved lateral and anterior teeth;
* no periodontal treatment in the last 12 months;
* intermediate or advanced periodontitis (Stage II / III / IV)
* in each quadrant at least three teeth with PPD>5 mm after initial treatment (scaling, motivation, instruction)

Exclusion Criteria:

* antibiotic therapy in the last 6 months;
* smoking;
* systemic diseases affecting periodontal tissues;
* pregnancy or lactation;
* orthodontic treatment;
* tooth mobility II / III degree;
* involvement of third degree furcations according to Hamp classification;
* endodontic issues

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | 0 (before), 3 and 6 months after SRP
  Distance from the gingival margin to the bottom of the gingival sulcus
Clinical attachment level (CAL) | 0 (before), 3 and 6 months after SRP
  Distance from the cementoenamel junction to the bottom of the gingival sulcus
Bleeding on probing (BoP) | 0 (before), 3 and 6 months after SRP
  Percentage of sites with bleeding provoked by applying a probe to the bottom of a sulcus/pocket.
Plaque index (PI) | 0 (before), 3 and 6 months after SRP
  Percentage of sites with plaque

SECONDARY OUTCOMES:
Width of keratinized tissue (KTW) | 0 (before), 3 and 6 months after SRP
  Distance between the most apical point of gingival margin and the mucogingival junction
Gingival thickness (GT) | 0 (before), 3 and 6 months after SRP
  Thickness of the gingiva measured 2 mm apical to the gingival margin

OTHER OUTCOMES:
Subgingival plaque pathogens (Aa, Pg, Td) levels | 0 (before) and 6 months after SRP
  Levels of periodontal pathogens (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Treponema denticola) measured with real-time polymerase chain reaction (RT-PCR) test; data presented as number of bacteria of these species and percentage of total bacteria found in a sample; sample taken from the deepest pocket on each side.
Gingival crevicular fluid levels of cytokines | 0 (before), 3 and 6 months after SRP
  Levels of (IL - interleukin) IL-1β, IL-6, IL-8, IL-10 and interferon-gamma in gingival crevicular fluid presented as pg/ml; sample taken from the deepest pocket on each side.

CONTACTS AND LOCATIONS:
Overall Officials: Bartlomiej Górski, PhD, Principal Investigator — Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw
Locations (1):
- Department of Periodontology and Oral Mucosa Diseases, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland